CLINICAL TRIAL: NCT02281617
Title: Smart-device Apps as Memory Aids
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: Maudsley Charity (Unknown)
Responsible Party: Sponsor
Other Study IDs: 139664
Record Dates: First submitted 2014-10-28; First posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Memory Disorders
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Smart-device apps as memory aids — Patients will be taught to use software running on smartphones and smart tablets to help compensate for memory difficulties

SUMMARY:
Patients experience problems with their memories from a variety of causes. There has been much work showing that the use of low tech devices, such as notebooks or diaries, can help patients remain independent. More recently, the use of electronic devices, such as digital voice recorders or pagers, has proved equally beneficial. Many of functions of memory aids could potentially be carried out by a smartphone or tablet using inbuilt functions such as a calendar or maps, as well as through downloadable apps, such as medication reminders. The investigators have surveyed the investigators patients to show that many of them already own smartphones and this number has dramatically increased in the last year. This project aims to investigate the feasibility and efficacy of using smartphone and tablet apps as memory aids in a clinical setting.

DETAILED DESCRIPTION:
Purpose and design

This study will trial the use of smartphones and apps as memory aids with patients who have memory problems. There have been some case study reports in the literature but the investigators would like to use this study to investigate how feasible it is to offer these kinds of support within an NHS memory aids service.

Recruitment

Patients (and their relatives/carers, where relevant)will be recruited from those already referred to the Memory Aids Service run within the Neuropsychiatry and Memory Disorders Clinic at St Thomas's Hospital, within the South London and Maudsley NHS Foundation Trust. It is made clear in the Participant Information Sheet (one for patients and one for relatives/carers) that participation is voluntary and if patients do not want to take part, they will still receive personalised help and advice in the Memory Aids Service.

Inclusion/Exclusion

This project will be offered to patients who own their own smartphone; the project is unable to support costs of buying smartphones for patients and paying for any data usage. Patients who do not have smartphones will still receive memory aids support, but instead will receive help as is standardly given using other memory aids.Patients will be excluded if they do not have adequate levels of English or motor skills to use the apps.

Consent

Patients will be identified as possible participants during their routine memory aids assessment clinic visit by a member of the clinical care team. Only those with capacity to consent will be invited to take part. Those interested in taking part will be given a patient information sheet at the end of their assessment appointment (as will their relatives/carers where relevant) and the study will be briefly explained orally. Patients (and their relatives/carers) who do decide to participate will sign the consent form at the beginning of their next Memory Aids appointment and it will be stressed that participation is voluntary and they can withdraw at any time.

Confidentiality

Access to clinical data (pre- and post- intervention memory, mood, functioning, goal and carer stress scores, neuropsychological test scores and interview transcripts) will be restricted to those in the clinical care team until data is fully anonymised. Patients will be asked for consent for their data to be used for the study and a specific point on the informed consent form should be initialled to allow this.

Risks, burdens and benefits

The investigators hope that patients will find benefits in using smartphones as memory aids. The investigators will pay for any apps that are selected to use with them and offer instructions. Use of electronic aids and alarms on phones is well practised within the existing memory aids service. This project adds a semi-structured interview and follow-up phone call and therefore a limited burden for research participants and in some cases their relatives/carers. Since the intervention is non-invasive, the risk to participants is very low.

ELIGIBILITY:
Inclusion Criteria:

* Subjective memory problems
* Fluent English
* Owns a smartphone or tablet
* sufficient motor skills to operate the smartphone or tablet
* sufficient eyesight to see the smartphone or tablet

Exclusion Criteria:

-

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults attending an NHS memory clinic with fluent English and in possession of a smart-phone or tablet
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Prospective and Retrospective Memory Questionnaire PRMQ | End of intervention, on average 2 months
  Subjective memory questionnaire
Meta-memory questionnaire MMQ | End of intervention, on average 2 months
  Questionnaire about beliefs about memory, problems and strategies
Hospital Anxiety and Depression Inventory HADS | End of intervention, on average 2 months
  Questionnaire about anxiety and depression
Revised carer stress index | End of intervention, on average 2 months
  Questionnaire about carer stress
Semi-structured interview | End of intervention, on average 2 months
  Semi-structured interview about usability and usefulness of memory aid apps
Brief phone call | 1 year post treatment
  Brief phone call to ask which apps are still being used

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Liebscher, MA, Study Director — South London and Maudsley NHS Foundation Trust

REFERENCES:
- [Background] Migo EM, Haynes BI, Harris L, Friedner K, Humphreys K, Kopelman MD. mHealth and memory aids: levels of smartphone ownership in patients. J Ment Health. 2015;24(5):266-70. doi: 10.3109/09638237.2014.951479. Epub 2014 Sep 4. PMID 25188922